CLINICAL TRIAL: NCT03188783
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GDC-0853 in Healthy Japanese and Caucasian Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GDC-0853 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP39851
Record Dates: First submitted 2017-06-14; First posted 2017-06-15 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — fenebrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: GDC-0853 Low Dose (Experimental): Japanese subjects will receive a single low dose of GDC-0853 or matching placebo by mouth.
  Interventions: Drug: GDC-0853; Drug: Placebo
- Cohort 2: GDC-0853 Intermediate Dose (Experimental): Japanese subjects will receive a single intermediate dose of GDC-0853 or matching placebo by mouth. Subsequently, participants will receive twice-daily intermediate doses of GDC-0853 or matching placebo by mouth for 4 days followed by a single intermediate dose of GDC-0853 or matching placebo by mouth.
  Interventions: Drug: GDC-0853; Drug: Placebo
- Cohort 3: GDC-0853 Intermediate Dose (Experimental): Caucasian subjects will receive a single intermediate dose of GDC-0853 or matching placebo by mouth. Subsequently, participants will receive twice-daily intermediate doses of GDC-0853 or matching placebo by mouth for 4 days followed by a single intermediate dose of GDC-0853 or matching placebo by mouth.
  Interventions: Drug: GDC-0853; Drug: Placebo
- Cohort 4: GDC-0853 Low Dose (Experimental): Japanese subjects will receive a single high dose of GDC-0853 or matching placebo by mouth.
  Interventions: Drug: GDC-0853; Drug: Placebo

INTERVENTIONS:
Drug: GDC-0853 — GDC-0853 tablets orally, either a single dose or twice-daily.
Drug: Placebo — GDC-0853 matching placebo tablets orally, either a single dose or twice-daily.

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics of single and multiple oral doses of GDC-0853 in healthy Japanese and Caucasian subjects.

DETAILED DESCRIPTION:
This study will be a randomized, placebo-controlled, double-blind, single and multiple dose study. Approximately 32 healthy subjects will be enrolled in 4 discrete cohorts with 8 subjects per cohort.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects must have both Japanese parents and all grandparents who were born in a Japanese country of origin
* Caucasian subjects must have 4 Caucasian grandparents (Hispanics of white race can be considered Caucasians)
* Within body mass index range of 18 to 31 kilograms per square meter, inclusive
* Females will be non-pregnant, non-lactating, and either postmenopausal or surgically sterile
* Males will either be sterile or agree to use an approved method of contraception

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic/immunologic/immunodeficiency, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the investigator)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* Participation in any other investigational study drug trial in which receipt of any investigational study drug occurred within 30 days or 5 half-lives, whichever is longer, prior to check in
* History of malignancy, except for appropriately treated carcinoma in situ of the cervix or non-melanoma skin carcinoma with 3-year disease-free follow up
* Any acute or chronic condition or any other reason that, in the opinion of the investigator, would limit the participant's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Cohorts 1 and 4: up to Day 29; Cohorts 2 and 3: up to Day 36
  An AE is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. Preexisting conditions which worsen during a study are also considered as adverse events. A SAE is any untoward medical occurrence that at any dose: results in death, or is life-threatening, or requires inpatient hospitalization or prolongation of existing hospitalization, or results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. The term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event, not an event which hypothetically might have caused death if it were more severe.
Number of Participants with Clinical Significant Change in Vital Sign, Physical Examination Findings, Clinical Laboratory Results and Electrocardiograms (ECGs) | Cohorts 1 and 4: up to Day 29; Cohorts 2 and 3: up to Day 36
  Number of participants with clinical significant change in vital sign, physical examination findings, clinical laboratory results and electrocardiograms (ECGs) will be reported.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of GDC-0853 | Predose and up to 72 hours postdose
  Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time 0 to 48 Hours Post-dose (AUC0-48) of GDC-0853 | Predose and up to 72 hours postdose
  Area under the concentration-time curve from Hour 0 to 48 hours postdose, calculated using the linear trapezoidal rule for increasing concentrations and the logarithmic rule for decreasing concentrations.
Area under the plasma concentration-time curve from time zero to time tau over the dosing interval (AUC0-tau) | Predose and up to 72 hours postdose
  Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States